CLINICAL TRIAL: NCT02856308
Title: Safety and Efficacy Evaluation of Hairstetics Hair Implant in Subjects Affected With Hair Loss - a Clinical Study
Brief Title: Hairstetics Hair Implant Device Safety and Efficacy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hairstetics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HET-03
Record Dates: First submitted 2016-07-07; First posted 2016-08-04 (Estimated); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: Alopecia
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hairstetics hair implant device (Experimental): Subjects will undergo the Hairstetics prosthetic hair implantation starting with a test of up to 100 fibers and up to 2 additional implantation sessions with up to 1500 fibers overall per subject. The implantation will be carried out according to the device IFU.
  Interventions: Device: Hairstetics hair implant device

INTERVENTIONS:
Device: Hairstetics hair implant device

SUMMARY:
This is a prospective, single-arm, multi-center, international, open-label, non-randomized, clinical study.

The aim of the study is to assess the safety and efficacy of the use of the Hairstetics hair implant device in subjects affected with hair loss.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥ 19 years old.
2. Subject has hair loss and has chosen to undergo synthetic hair implantation.
3. Subject has mental capacity to understand study guidelines and requirements (to maintain scalp hygiene, use of shampoo, delicate combing, etc.).
4. Subject has been evaluated by the investigator to have a scalp condition in the planned area of implantation that is acceptable for entering the study and currently is NOT suffering from skin problems at planned implantation site or elsewhere that might affect the procedure and/or success as clinically evaluated by the investigator.
5. Subject has Good general health.
6. Woman of child bearing potential must have a negative pregnancy test.
7. Subject willing to sign a written informed consent form (ICF) and the post implantation maintenance protocol.

Exclusion Criteria:

1. Previous synthetic hair implantation or hair transplantation in the past 6 months.
2. Currently suffering from skin problems at planned implantation site or elsewhere that might affect the procedure and/or success as clinically evaluated by the investigator.
3. Currently receiving or have within the past 3 months received radiation- and/or chemotherapy.
4. Currently using steroid product with Immunosuppressive treatment.
5. Impaired coagulation.
6. Serious illness that may affect subject compliance to protocol.
7. Subject is using illegal drugs.
8. Participating in other clinical study.
9. Known allergy or hypersensitivity to Nitinol or Nickel or Titanium
10. For woman: Pregnancy or breast feeding.
11. Known allergy or intolerance for the prescribed antibiotics and in such a case, a different antibiotics for which the subject is not allergic or intolerance to, will be prescribed

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-03; Primary Completion 2018-03 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Acceptable number, duration and severity of expected adverse device/procedure effects | 3 months following implantation

CONTACTS AND LOCATIONS:
Locations (8):
- France (3):
  - Cabinet du Dr G. Beilin, Paris
  - Cabinet médical du Dr Jack Smadja, Paris
  - Georges Mandel Office Surgery Clinic, Paris
- India (2):
  - Paras hospital, Gūrgaon
  - Fortis Hospital, New Delhi
- Romania (2):
  - Egoclinic, Bucharest
  - Metropolitan hospital, Bucharest
- Revere clinic, London, United Kingdom